CLINICAL TRIAL: NCT03889340
Title: Study of Brain Cools Device in Patients Resuscitated From Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Adam Frisch (Other)
Collaborators: BrainCool (Unknown)
Responsible Party: Sponsor-Investigator, Adam Frisch, Assistant Professor of Emergency Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: PRO18060375
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Arrest With Successful Resuscitation
Keywords: resuscitation; cardiac arrest; coma
MeSH Terms: conditions — Heart Arrest; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Phase 1 cohort: Subjects resuscitated from cardiac arrest will undergo cooling per standard of care with the IQool device.
  Interventions: Device: IQool

INTERVENTIONS:
Device: IQool — Subjects will undergo hypothermia therapy with the IQool system

SUMMARY:
This submission is a pilot in which the new IQool Warming System device will be used to maintain the temperature of adult patients in cardiac arrest within a range of within a range of 32°C to 38.5°C (89.6°F to 101.3°F). The IQool Warming System has received a 510 K Clearance by the FDA.

DETAILED DESCRIPTION:
Subjects will receive temperature management using the IQool. This is an FDA approved device. Managing temperature is part of standard care for this population and surface cooling is commonly employed.

The following phases will be conducted as standard of care, and will be reviewed for this study:

Induction phase: When a subject is included in the study, the IQool will be connected to the patient and activated. The induction period will continue until the patient has reached the upper limit of the target temperature range (defined as 0.5°C above the target temperature).

Maintenance phase: Set target temperature will be maintained for 24 hours. The maintenance phase begins when the subject temperature is within 0.5°C of goal temperature. The maintenance phase is completed 24 hours after first reaching below the upper limit of the target temperature range.

Rewarming phase: After 24 hours of maintenance, gradual rewarming at 0.25 °C/h will commence. When the subject reaches 37°C the TTM period is completed and the IQool will continue to provide fever control.

Post TTM fever control: The subject will be kept at a body temperature of 37°C until 72 hours after the cardiac arrest or earlier if the subject regains consciousness.

ELIGIBILITY:
Inclusion Criteria:

* In- or out-of-hospital cardiac arrest of all initial rhythms
* Adult patients (18 years of age and older)
* Unconscious on admission to hospital, defined as not following commands
* Indication for targeted temperature management

Exclusion Criteria:

* Pregnancy
* Prisoner
* Active do not resuscitate order
* Any patient not expected to survive 72 hours
* Skin infection
* Skin wound affecting site of temperature exchange pads

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be cardiac arrest patients that have been successfully resuscitated.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of hypothermia induction | Up to 12 hours
  Induction of hypothermia will occur at a rate of at least 1C/hr
Maintenance of hypothermia | 24 hours
  The IQool system will maintain temperature within 0.5C of goal temperature for 75% of the maintenance phase
Rewarming rate | Up to16 hours
  When rewarming, the IQool system will rewarm within 0.5C of the goal rate of rewarming

SECONDARY OUTCOMES:
Number of physicians that recommend the IQool system for temperature management | 72 hours
  Clinicians will be asked if they agree that the IQool system provides effective temperature management >90% of the time

CONTACTS AND LOCATIONS:
Overall Officials: Jon Rittenberger, MD, Principal Investigator — Associate Professor of Emergency Medicine, University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States